CLINICAL TRIAL: NCT00434083
Title: A Double-Blind Multicenter, Randomized, Placebo-Controlled Single Dose Study to Evaluate the Safety and Efficacy of Trexima in the Acute Treatment of Migrane Headaches
Brief Title: To Evaluate the Safety and Efficacy of Trexima in the Acute Treatment of Migrane Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT400-301
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Migraine Headaches
Keywords: TREXIMA; MIGRAINE HEADACHES; Subjects may be enrolled if they are 18-65 years of age, have a demonstrated history of migraine headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

INTERVENTIONS:
Drug: sumatriptan
Drug: naproxen sodium

SUMMARY:
* to demonstrate the superiority of Trexima (combination of sumatriptan as the succinate 85 mg and naproxen sodium 500 mg) versus placebo in the acute treatment of migraine
* to demonstrate the superiority of Trexima versus the individual components (sumatriptan as the succinate 85 mg and naproxen sodium 500 mg), and
* to evaluate the safety of the Trexima.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study if all of the following criteria apply:

1. Subject is a male or a female who is not pregnant or is not lactating. A female is eligible to enter and participate in this study if she is of

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant): or,
   * Child-bearing potential, has a negative pregnancy test (urine or serum) at screen, and employs one of the following acceptable measures of contraception:

     * Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug (a minimum of 24 hours); subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for randomized treatment; or
     * Female sterilization; or
     * Sterilization of male partner; or implants of levonorgestrel; or
     * Injectable progestogen; or
     * Oral contraceptive (combined or progestogen only); or
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or
     * Any other method with published data showing that the lowest expected failure rate for that method is less than 1% per year.
     * Barrier method only if used in combination with any of the above.
2. Subject is 18-65 years of age.
3. Subject's first migraine occurred prior to the age of 50 years.
4. Subject has at least a 6-month history of migraine with or without aura according to the International Headache Society criteria (see Appendix I).
5. Subject experienced an average migraine headache frequency of 2-6 moderate or severe attacks per month in the previous 3 months.
6. Subject is able to distinguish his/her migraine attacks as discrete from any other types of headaches.
7. Subject is willing and able to give written informed consent prior to entry into the study.

Exclusion Criteria:

* A subject will not be eligible for this study if any one or more of the following criteria apply:

  1. Subject has received another investigational drug within the 4 weeks preceding this study, subject was discontinued from the MT400-303 POZEN study, or subject was enrolled in this study or the MT400-302 POZEN study previously.
  2. Subject has any concurrent medical or psychiatric condition that may affect the interpretation of efficacy and/or safety data or which otherwise contraindicates participation in a clinical trial with a new chemical entity. This includes, but is not limited to, chronic unstable debilitating diseases such as HIV infection, multiple sclerosis, cancer, etc.
  3. Subject has a clinically significant disorder that, in the opinion of the investigator, would result in the subject's inability to understand and comply with the requirements of the study.
  4. Subject has a history, signs, or symptoms of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes or other significant underlying cardiovascular disease.
  5. Subject has a history of cardiac arrhythmias requiring medication or a history of a clinically significant electrocardiogram (ECG) abnormality that, in the investigator's opinion, contraindicates participation in this study.
  6. Subject has a history of cerebrovascular pathology including stroke and/or transient ischemic attacks.
  7. Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular disease, based on history or the presence of risk factors (e.g., hypertension, hypercholesterolemia, smoker, obesity, diabetes, strong family history of coronary artery disease, female with surgical or physiological menopause, or male over 40 years of age).
  8. Subject has evidence or history of ischemic abdominal syndromes, peripheral vascular disease, or Raynaud syndrome.
  9. Subject has uncontrolled hypertension at screening (sitting systolic pressure >160 millimeters of mercury [mmHg], diastolic pressure >95 mmHg).
  10. Subject has a history of epilepsy or conditions associated with a lowered seizure threshold.
  11. Subject has a history of basilar or hemiplegic migraine.
  12. Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study, or the subject has any other abnormal laboratory value of clinical significance for this study.
  13. Subject has a history of non-migraine (i.e., tension type, sinus, etc.) headache frequency greater than or equal to 15 days/month in each of the 3 months prior to screening.
  14. Subject has had >6 migraine attacks/month in either of the 2 months prior to screening.
  15. Subject is currently taking a monoamine oxidase inhibitor (MAOI), has taken an MAOI within the 2 weeks prior to screening, or plans to take an MAOI within 2 weeks after treatment.
  16. Subject is currently taking any anti-coagulant (e.g. warfarin) or NSAID (except doses of aspirin ≤ 325 mg per day, used for cardiovascular prophylaxis) on a regular basis.
  17. Subject is currently taking or has taken in the previous 3 months, a migraine prophylactic medication containing ergotamine, an ergot derivative (dihydroergotamine), or methysergide.
  18. Subject is currently taking or has taken in the previous 4 weeks, herbal preparations containing St. John's Wort (Hypericum perforatum).
  19. Subject has hypersensitivity, intolerance, or contraindication to the use of sumatriptan or naproxen sodium, any of its components, or any other 5-HT1 receptor agonist.
  20. Subject has history of allergic reactions to naproxen preparations, including subjects in whom aspirin or other NSAID drugs induce the syndrome of asthma, rhinitis, and nasal polyps.
  21. Subject is pregnant, actively trying to become pregnant, or breast-feeding.
  22. Subject is of childbearing potential and not using adequate contraceptive measures.
  23. Subject has a recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse (abuse) of ergotamines and/or narcotics to treat migraines. Ergotamine abuse is daily use for 14 consecutive days or intermittent consumption exceeding 10 mg per week for any two weeks.
  24. Subject has participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during the period of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2004-07; Study Completion 2005-01

PRIMARY OUTCOMES:
Trexima will be evaluated for efficacy as an acute treatment for migraine based on its superiority over placebo at 2 hours for: a) pain relief (no or mild pain), b) incidence of photophobia, c) incidence of phonophobia and d) incidence of nausea.

SECONDARY OUTCOMES:
a) sustained pain relief over 24 hours, b) sustained photophobia-free over 24 hours, c) sustained phonophobia-free over 24 hours, and d) sustained nausea-free over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: David Taylor, Study Director — POZEN
Locations (2):
- United States (2):
  - Pozen, Inc., Chapel Hill, North Carolina
  - Nashville Neuroscience Group, PC, Nashville, Tennessee

REFERENCES:
- [Derived] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970